CLINICAL TRIAL: NCT01267383
Title: Open Label, Balanced, Randomized, Two Treatment, Two Sequence, Two Period, Single-dose, Crossover Oral Bioequivalence Study of Sertraline Hydrochloride 100 mg Tablets (Dr. Reddy's Laboratories Limited, India) With the Reference Formulation ZOLOFT® 100 mg Tablet (Pfizer, USA)Under Fed Conditions in Healthy Human Adult Subjects.
Brief Title: Bioequivalence Study of Sertraline Hydrochloride Tablets 100 mg in Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sr. Director- Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06-VIN-102
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2012-01-11 (Estimated); Status verified 2012-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Sertraline; crossover
MeSH Terms: interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sertraline Hydrochloride tablets 100 mg (Experimental): Sertraline Hydrochloride tablets 100 mg of Dr.Reddy's Laboratories Limited
  Interventions: Drug: Sertraline
- Zoloft 100 mg Tablets (Active Comparator): Zoloft 100 mg Tablets of Pfizer
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — Sertraline Hydrochloride Tablets 100 mg
  Other Names: Zoloft

SUMMARY:
The objective of this study was to compare and evaluate the single-dose oral bioavailability of the test formulation of Sertraline Hydrochloride 100 mg tablets (Dr. Reddy's Laboratories Limited) with the reference formulation ZOLOFT® 100 mg Tablet (Pfizer)under fed conditions in healthy adult human subjects.

DETAILED DESCRIPTION:
Open Label, Balanced, Randomized, Two Treatment, Two Sequence, Two Period, Single-dose, Crossover, Oral Bioequivalence Study of Sertraline Hydrochloride 100 mg Tablets (Dr. Reddy's Laboratories Limited, India) With the Reference Formulation ZOLOFT® 100 mg Tablet (Pfizer, USA)Under Fed Conditions in Healthy Human Adult Subjects. 32 healthy, adult, human male subjects were enrolled in the study and all the subjected completed all the periods.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy human subjects ages 18 and 45 years (including both).
2. Subjects weight within the normal range according to normal values for the body mass index (18.5 to 24.9 kg/m2) with minimum of 50 kg weight.
3. Subjects with normal health as determined by personal medical history, clinical examination and laboratory examinations within the clinically acceptable normal rane.
4. Subjects having normal 12-lead electrocardiogram (ECG)
5. Subjects having normal chest X-Ray (P/A view)
6. Subjects having negative urine screen for drugs of abuse(including amphetamines, barbiturates, benzodiazepines, marijuana, cocaine, and morphine).
7. Subjects having negative alcohol breath test
8. Subjects willing to adhere to the protocol requirements and to provide written informed consent.

For Female Subjects:

1. Female of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies,diaphragm, intrauterine devise(IUD) or abstinence, or
2. Postmenopausal for at least 1 year or
3. Surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject.

Exclusion Criteria:

1. Hypersensitivity to sertraline hydrochloride or related class of drugs.
2. History or presence of significant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, endocrine, immunological, dermatological neurological or psychiatric disease or disorder.
3. Any treatment which could bring about induction or inhibition of hepatic microsomal enzyme system within 1 month of the study starting.
4. History or presence of significant alcoholism or drug abuse in the past one year.
5. History or presence of significant smoking (more than 10 cigarettes day) or consumption of tobacco products.
6. History or presence of significant asthma, urticaria or other allergic reactions.
7. History or presence of significant gastric and/or duodenal ulceration.
8. History or presence of significant thyroid disease, adrenal dysfunction, organic intracranial lesion such as pituitary tumor.
9. History or presence of cancer
10. History or presence of significant easy bruising or bleeding
11. History or presence of significant recent trauma
12. Subjects who have been on an abnormal diet(for whatever reason) during the four weeks preceding the study.
13. Difficulty with donating blood
14. Difficulty in swallowing solids like tablets or capsules
15. Systolic blood pressure less than 100 mm Hg or more than 140 mm Hg
16. Diastolic blood pressure less than 60 mm Hg or more than 90 mm Hg.
17. Pulse rate less than 50/minute or more than 100/minute
18. Oral temperature less than 95ºF or more than 98.6ºF.
19. Respiratory rate less than 12/minute or more than 20/minute
20. Use of any prescribed medication during last two weeks or OTC medical products during the last week prior to initiation or study
21. Major illness during 3 months before screening
22. Participation in a drug research study within past 3 months
23. Donation of blood in the past 3 months before screening.

For Female Subjects:

Female subjects who are pregnant or who are able (women with child bearing potential) to become pregnant during the study were not allowed to participate.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-09; Primary Completion 2006-09 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Damesh Domadia, MBBS, M.D, Principal Investigator — Veeda Clinical Research (P) Ltd
Locations (1):
- Veeda Clinical Research (P) Ltd, Ambawadi, Ahmedabad, India